CLINICAL TRIAL: NCT04857190
Title: Parker Flex-it Directional Stylet Versus Conventional Malleable Stylet in Elective Orotracheal Intubation Using a Fiber-optic Laryngoscope
Brief Title: Parker Flex-it Stylet Versus Malleable Stylet in Orotracheal Intubation Using a Fiber-optic Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DTH: 21001
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-04

CONDITIONS: Orotracheal Intubation
Keywords: Conventional Malleable Stylet; Orotracheal Intubation; Parker Flex-it Directional Stylet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DS (n=40) (Active Comparator): Parker Flex-it Directional Stylet group
  Interventions: Device: Parker Flex-it Directional Stylet
- Group MS (n=40) (Active Comparator): Conventional Malleable Stylet group
  Interventions: Device: Conventional Malleable Stylet

INTERVENTIONS:
Device: Parker Flex-it Directional Stylet — Parker Flex-it Directional Stylet
  Arms: Group DS (n=40)
Device: Conventional Malleable Stylet — Conventional Malleable Stylet
  Arms: Group MS (n=40)

SUMMARY:
Objectives: To compare the safety and efficacy of Parker flex-it directional stylet (PFDS) versus conventional malleable stylet (CMS) in orotracheal intubation (OTI) using fiber-optic Macintosh laryngoscope.

Background: OTI is used in general anesthesia for anesthetic delivery and ventilation of patients. OTI delay or failure may adversely affect patient outcomes, therefore, anesthetists with sufficient clinical experience and skill should perform OTI. However, in emergency situations, experienced anesthetists may not be available, and the patient may have a high Cormack-Lehane grade. A stylet is commonly used in the emergency department to aid insertion of the endotracheal tube during direct laryngoscopy.

Patients and Methods: This was a prospective, randomized, double-blind clinical trial; carried out on 80 patients requiring OTI under general anesthesia at our hospital. Patients were randomly allocated into two equal groups; group DS, intubated using PFDS, and group MS, intubated using CMS.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 60 years
* Body Mass Index (BMI) < 35
* Mallampati classification ≤ II

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status > II
* Age < 21 years or > 60 years
* Body Mass Index (BMI) ≥ 35
* Mallampati classification > II
* Pregnant women
* Anticipated difficult airway
* Need for rapid sequence induction
* Increased risk of gastric aspiration such as gastroesophageal reflux
* Edentulous patients, Loose teeth
* Known pathology, trauma, or previous surgery to the mouth, pharynx, larynx, or cervical spine
* History of; Dysrhythmia, Hypertension, Ischemic heart disease, Hyperthyroidism, DM

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Mean and Standard deviation of Time required for orotracheal intubation (seconds) (mean±SD) | 2 minutes after inserting the blade of the laryngoscope in the mouth
  Time interval from holding the endotracheal tube by the anesthetist till removal of the stylet from the endotracheal tube by the anesthetist

SECONDARY OUTCOMES:
Mean and Standard deviation of Total time required for orotracheal intubation (seconds) (mean±SD) | 2 minutes after inserting the blade of the laryngoscope in the mouth
  Time interval from inserting the blade of the laryngoscope into the patient's mouth till the appearance of end-tidal carbon dioxide curve of at least 30 mmHg on the anesthesia monitor after insertion of the endotracheal tube
Mean and Standard deviation of Number of intubation attempts (mean±SD) | 2 minutes after inserting the blade of the laryngoscope in the mouth
  An attempt is the act of inserting and removing the blade of the laryngoscope from the mouth
Number of participants and Rate of Successful intubation from the first-attempt | 2 minutes after inserting the blade of the laryngoscope in the mouth
  First-attempt intubation success rate
Number of participants and Rate of Use of external laryngeal manipulation | 2 minutes after inserting the blade of the laryngoscope in the mouth
  Number of participants and Rate of Use of external laryngeal manipulation
Mean and Standard deviation of Heart rate (beat/min.)(mean±SD) | 2 minutes after inserting the blade of the laryngoscope in the mouth
  Before, after induction, and 2 minutes after inserting the blade of the laryngoscope in the mouth
Mean and Standard deviation of Oxygen Saturation (%)(mean±SD) | 2 minutes after inserting the blade of the laryngoscope in the mouth
  Before, after induction, and 2 minutes after inserting the blade of the laryngoscope in the mouth
Mean and Standard deviation of Blood Pressure (mmHg)(mean±SD) | 2 minutes after inserting the blade of the laryngoscope in the mouth
  Before, after induction, and 2 minutes after inserting the blade of the laryngoscope in the mouth
Number of participants and Rate of Procedure-related complications | 5 minutes after the end of the procedure
  Number of participants and Rate of: Tachycardia, Dysrhythmia, Hypoxemia, Hypertension, Laryngospasm, Bronchospasm, Oropharyngeal trauma

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt